CLINICAL TRIAL: NCT05599711
Title: Testing the Efficacy of an Adapted Family-Centered Autism Transition Intervention in a Safety Net Hospital Setting
Brief Title: Transitioning Together Boston
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Deborah Munroe Noonan Memorial Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-43047
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Autism or Autistic Traits; Family Relations
Keywords: Multi-family group intervention sessions; Psychoeducational autism transition-to-adulthood; Problem-solving education; Quality of life of autistic youth; Goal attainment; Parent-youth dyad
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitioning Together (Experimental): Participants in this arm will receive the Transitioning Together intervention in English or Spanish either at BMC, at BMC's Supporting Parents & Resilient Kids (SPARK) Center or on BMC Zoom.
  Interventions: Behavioral: Transitioning Together (TT) / Juntos en la Transicion (JET)
- Usual Care (Active Comparator): Participants in this arm will receive a referral to usual transition-related care through the BMC Developmental and Behavioral Pediatrics (DBP) clinic/the BMC Autism Program.
  Interventions: Behavioral: Usual autism transition care

INTERVENTIONS:
Behavioral: Transitioning Together (TT) / Juntos en la Transicion (JET) — 1. One individual family joining session when each family dyad meets with group therapists to establish rapport and share their own unique family's background, goals, and supports.
  2. A series of four 2.5-hour multi-family group psychoeducation intervention sessions focused on problem-solving education and psychoeducational autism transition-to-adulthood content which can include independence in adulthood, community involvement, guardianship and legal issues, employment and education, health and well-being.
  Arms: Transitioning Together
Behavioral: Usual autism transition care — An expedited referral will be made for participants to establish care with a BMC Autism Program Transition/Resource Specialist. Data will be abstracted from the electronic medical record on how many visits each family completes with a BMC Autism Program Transition/Resource Specialist or other BMC Developmental and Behavioral Pediatrics provider throughout the study period.
  Arms: Usual Care

SUMMARY:
A randomized controlled trial will be conducted to determine the effects of an adapted family-centered autism transition intervention called Transitioning Together/Juntos en la Transición on meaningful outcomes for families. The study will occur in a safety net hospital setting. The adapted version of this multi-family group psychoeducation intervention is delivered across one individual family joining session and four 2.5 hour multi-family group sessions. The parent and youth groups are held in separately, at the same time.

DETAILED DESCRIPTION:
Objective 1: The investigators will test the efficacy of the adapted version of Transitioning Together on youth quality of life and progress toward individual transition goals. 128 English and/or Spanish speaking families of youth ages 14-21 years will be enrolled in the study. The primary enrollment site is Boston Medical Center (BMC), an urban safety net hospital where patients predominantly (>75%) from low-income households are served. The effects of Transitioning Together will be compared to a usual care control condition with a referral to the Transition Specialist within BMC's Developmental and Behavioral Pediatrics clinic. Youth quality of life and progress toward individual transition goals will be compared from baseline and three-to-six months following randomization. The investigators hypothesize that Transitioning Together will have a significant positive effect on youth quality of life and goal attainment across the two time points.

Objective 2: Additional standardized assessments will be administered to the 128 parents and the 128 autistic youth, to examine the effects of Transitioning Together compared to the control condition on: the broader family unit's well-being, empowerment, coping skills, social support, transition readiness, and family climate. The investigators will explore whether these factors act to mediate or moderate primary or secondary study outcomes (youth quality of life and progress toward individual transition goals). These putative mediators and moderators will be assessed at the baseline and 3-to 6-months following randomization.

ELIGIBILITY:
Inclusion Criteria for youth:

* Age 14 to 21 years old
* Be enrolled in high school or a specialized continued schooling program for youth ages 18 to 21.
* Has been seen at BMC at least once since 2015
* Confirmation of the autism diagnosis
* Currently live at home with a parent/legal guardian
* A parent/legal guardian who meets the below criteria

Inclusion Criteria for parents:

* Age at least 21 years old
* Parent/legal guardian of a youth who meets the youth criteria
* Parent/legal guardian is comfortable reading, writing, speaking, and listening in English and/or Spanish

Exclusion Criteria:

* A primary home language for the family is not English or Spanish (the intervention and assessments are only available in English and Spanish)
* The autistic youth currently resides independently, in supported housing, or with a foster family or other Department of Children and Families (DCF) placement
* Either the youth or their parent/guardian chooses not to participate in the study (one cannot participate without the other)

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life of autistic youth | Baseline, 3-12 months
  The Global Health, Emotional Distress, Subjective Well-Being, and Relationships sub scales of the NIH Patient-Reported Outcomes Measurement Information Systems (PROMIS) will be administered via parent proxy (and youth self-report when appropriate) to asses the quality of life for autistic youth. Item scores can range from 1 to 5 and higher scores are associated with a higher quality of life.
Change in transition-related goal attainment | Baseline, 3-12 months
  The Goal Attainment Scaling will be administered to asses transition-related goal attainment. It is a valid and reliable technique to benchmark success in meeting individualized goals. Scores can range from 0 to 4 and higher scores are associated with better goal attainment.
Change in youth problem behaviors | Baseline, 3-12 months
  The Scales of Independent Behavior-Revised Problem Behavior Scale will be administered to assess frequency and severity of problem behaviors in youth. It is a parent-report questionnaire. For problem behaviors that occurred, items scores can range from 1 to 5 for frequency and severity, with a higher score associated with higher frequency and higher severity of the problem behavior.

SECONDARY OUTCOMES:
Change in family empowerment | Baseline, 3-12 months
  The Family Empowerment Scale will be administered to asses family empowerment. It is a self-report scale that measures empowerment in families with children who have emotional or behavioral disorders and has robust psychometric properties. Item scores can range from 1 to 5 and higher scores are associated with more family empowerment.
Change in coping | Baseline, 3-12 months
  The Brief Coping Orientation to Problems Experienced Inventory (COPE) will be administered to asses family coping skills. It is a self-report questionnaire that measures adaptive and maladaptive coping responses to adversity, validated in health-care settings. Item scores can range from 1 to 4 and higher/lower subscale scores are associated with a higher level of the coping style measured in that subscale.
Change in social support | Baseline, 3-12 months
  The Medical Outcomes Study (MOS) Social Support Survey will be administered to asses social support. It is a self-report questionnaire that measures the availability of other people to provide social support through emotional, informational, tangible, affectionate, and social dimensions. Item scores can range from 1 to 5 and higher scores are associated with more social support.
Change in perceived burden | Baseline, 3-12 months
  The Zarit Burden Interview will be administered to asses perceived burden related to taking care of another person. It is a self-report questionnaire. Item scores can range from 0 to 4 and higher scores are associated with more perceived burden.
Change in parental well-being | Baseline, 3-12 months
  The Generalized Anxiety Screener and the Patient Health Questionnaire will be administered to asses parental well-being - specifically anxiety and depression symptoms. Both measures are self-report questionnaires. It is a self-report questionnaire. On the both measures, item scores range from 0 to 3 and higher scores are associated with higher severity of symptoms.
Change in family climate | Baseline, 3-12 months
  The Five-Minute Speech Sample and the Happy Proud Scale will be administered to asses family climate. The Five Minute Speech Sample is a 5-minute sample of a caregiver speaking about their relationship with their child that is scored to measure caregivers' expressed emotion regarding a relative with a mental health condition. The Happy Proud Scale measures parent and youth feelings of pride and happiness with regard to the things the youth does. Item scores range from 0 to 4 with higher scores associated with higher feelings of pride and happiness.
Change in transition readiness | Baseline, 3-12 months
  The Transition Readiness Scale will be used to assess youth readiness for the transition to adulthood. It is a parent proxy and youth self-report questionnaire. Item scores range from 1 to 4. Higher scores are associated with higher transition readiness.
  Additionally, the Waisman Activities of Daily Living Scale will be used to assess the level of independent aspect of transition readiness. It is a parent proxy report questionnaire. Item scores range from 0 to 2. Higher scores are associated with higher independence in performing tasks on one's own.

OTHER OUTCOMES:
Intervention acceptability, appropriateness, and feasibility | 3-12 months
  The Acceptability of Intervention Measure, the Intervention Appropriateness Measure, and the Feasibility of Intervention measure will be used to assess perceptions of intervention acceptability, appropriateness, and feasibility among participants who received the Transitioning Together intervention. These are each brief self-report questionnaires. Item scores range from 1 to 4. Higher scores are associated with higher perceptions of intervention acceptability, appropriateness, and feasibility.
Intervention Satisfaction | At the conclusion of each group session
  Participants receiving the Transitioning Together intervention will rate their satisfaction with each session on a self-reported satisfaction survey. Item scores range from 1 to 5. Higher scores are associated with a higher level of satisfaction.
Intervention Engagement | At the conclusion of each group session
  Facilitators will rate participant engagement level after each Transitioning Together session to measure their level of engagement. Scores range from 1 to 5. Higher scores are associated with a higher level of engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn L Kuhn, PhD, Principal Investigator — Emory School of Medicine; Mei Elansary, MD, Principal Investigator — Boston Medical Center, Pediatrics
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.